CLINICAL TRIAL: NCT05385029
Title: Thyroid Function Tests in Infants of COVID-19 Positive Pregnant Mothers
Brief Title: Fetal and Neonatal Thyroid in Pregnancies With Severe Acute Respiratory Syndrome Coronavirus 2 ( SARS- COV2 ) COVID-19
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: OMER B ABDELBASIT (Other)
Responsible Party: Sponsor-Investigator, OMER B ABDELBASIT, Consultant Neonatologist- Chief of Neonatal Intensive Care Unit ( NICU ), Security Forces Hospital
Organization: Security Forces Hospital (Other)
Other Study IDs: SecurityFH OABDELBASIT
Record Dates: First submitted 2022-05-10; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Thyroid Dysfunction; Hypothyroidism; Hyperthyroidism
Keywords: TSH Thyroid- Stimulating Hormone; FT4 Free Thyroxine; COVID-19 Corona Virus Disease; PCR Polymerase Chain Reaction; SARS COV2 Severe Acute Respiratory Syndrome; mIU milli-International Unit
MeSH Terms: conditions — Hypothyroidism; Hyperthyroidism | interventions — Thyroxine; Carbimazole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thyroid functions in neonates born to COVID 19 positive mothers: thyroid hormone or antithyroid drugs
  Interventions: Drug: Thyroxine
- Neonates born to mothers without COVID 19 infection: Thyroid drugs if indicated
  Interventions: Drug: Thyroxine

INTERVENTIONS:
Drug: Thyroxine — treatment for hypothyroidism or hyperthyroidism
  Other Names: Carbimazole

SUMMARY:
The thyroid gland has been shown to be a common target for COVID 19 virus. Babies born to mothers positive for COVID 19 infections were noticed to have elevated thyroid stimulating hormone ( TSH ) levels on screening. Thyroid function tests were monitored in these babies to determine presence of temporary or permanent thyroid disorders following COVID 19 infections during pregnancy.

DETAILED DESCRIPTION:
TSH estimation is carried out in all newborn babies in Saudi Arabia as a screening test for hypothyroidism. The first babies who were born to COVID 19 positive mothers were noticed to have significantly abnormal high TSH values. All the data and studies on the effect of COVID 19 on thyroid gland are from adult literature. Hence with these results of TSH in the the newborns we designed this observational study to monitor the thyroid functions in infants of COVID 19 positive mothers born in our hospital. The study confirmed presence of abnormal TSH and free thyroxine in these babies at birth and these babies were followed further after that for evidence of thyroid disorders.Results of thyroid functions in the babies who born in the same period of the study to mothers without COVID 19 infection were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* All newborns

Exclusion Criteria:

* Babies with congenital malformations

Age Groups: Child, Adult, Older Adult
Study Population: All newborn babies delivered in Security Forces Hospital
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Presence of Thyroid Dysfunction as Hypothyroidism or Hyperthyroidism | First measurement of TSH at birth to 24 hours. Then repeat TSH and FT4 after 48-72 hours
  Measurement of TSH values in mIU/l and FT4 values in pool/l. In our Hospital laboratory a TSH value above 35 mIU/l is suggestive of primary hypothyroidism while an FT4 level below 12 pmol/l would confirm the diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Security Forces Hospital, Riyadh, Central, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
After statistical analysis all data will be shared for discussion and final approval
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 3 moths